CLINICAL TRIAL: NCT02034695
Title: Evaluation of Quality of Care - Risk Assessment Management Programme, HA
Acronym: QoC RAMP
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Clinical Professor, The University of Hong Kong
Other Study IDs: HKCTR-1186
Record Dates: First submitted 2013-08-28; First posted 2014-01-13 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RAMP and Non-RAMP

SUMMARY:
Diabetes mellitus (DM) is one of the major cause of morbidity and among the top 10 causes of deaths in Hong Kong in 2008 (Department of Health 2009). The Hospital Authority (HA) has initiated service improvement through introducing the risk assessment and management programme (RAMP) to improve the quality of care (QOC) for DM patients in general outpatient clinics (GOPC). The evaluation on the QOC is an essential part of the programme in order to inform future policy. The Department of Family Medicine and Primary Care (FMPC) of the University of Hong Kong (HKU) has been appointed by the HA to carry out the evaluation of the QOC of the programme.

The Action Learning and Audit Spiral methodologies to measure whether the target standard of care intended by the RAMP programme is achieved. Each RAMP participating clinic and hospital will be invited to complete a structured evaluation questionnaire. The data of all patients who have enrolled into the RAMP for more than one year will be included in the evaluation on the process and outcomes of care.

One thousand two hundred and forty-eight age and disease matched control patients who have not been enrolled into the RAMP programme will be selected for the comparison in the outcomes of care. A hundred and thirty participants will be followed up by telephone to evaluate the effect of the programme in quality of life (QOL), patient enablement, and global rating of change in health condition at baseline and 6 months after enrolment. Data on the process of care will be retrieved from the HA medical records.

Main Outcome Measures: The primary outcomes are the proportion of participants who have received the criterion process of care, and achieved the target HbA1c and blood pressure levels.

Data Analysis: Descriptive statistics on proportions of centers or subjects meeting the QOC criteria will be calculated. The changes in the clinical and patient reported outcomes of RAMP subjects will be compared at 12, 24, 36 and 48 months will be compared by paired sample t-test. The clinical outcomes between RAMP subjects and control group will be compared by independent sample t-test or Chi-square test.

Results: The QOC of the RAMP programme will be determined. Areas of deficiency and possible areas for quality enhancement will be identified.

Conclusion: The results of this study will provide empirical evidence on whether the HA's RAMP programme can achieve improvement in QOC for DM patients. The information will be used to guide service planning and policy decision making.

ELIGIBILITY:
Inclusion Criteria:

* Patients with DM who are mostly independent in their activities of daily living and being followed up at GOPC regularly will be recruited.

Exclusion Criteria:

* Patients will be excluded if they are unable to understand or communicate in Chinese language, or refuse to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with DM who are mostly independent in their activities of daily living and being followed up at GOPC regularly will be recruited. All enrolled patients will undergo a comprehensive risk assessment and screening for complications, who will then be assigned to receive appropriate interventions and education from multi-disciplinary healthcare professionals according to their risk level. Low risk patients will continue with the usual GOPC follow up, medium risk patients will be given additional intervention by an advanced practice nurse (APN), and high risk patients will be given additional intervention by an APN and an associate consultant (AC) in family medicine (FM).
Sampling Method: Probability Sample
Enrollment: 2496 (Actual)
Dates: Start 2010-09; Primary Completion 2016-09 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The proportion of clinics that have satisfied each of the structure criteria | Five years
  Interim analysis will evaluate the period from August, 2009 to December, 2010; to December, 2011; to December, 2012; to December, 2013. Final analysis will evaluate the period from August, 2009 to December, 2014.
The proportion of patients who have complied with the criterion process of care. | Five years
  Interim analysis will evaluate the period from August, 2009 to June, 2011; to December, 2011; to December, 2012; to December, 2013. Final analysis will evaluate the period from August, 2009 to December, 2014.
The proportion of patients who have achieved a HbA1c level <7%. | Five years
  Interim analysis will evaluate the period from August, 2009 to June, 2011; to December, 2011; to December, 2012; to December, 2013. Final analysis will evaluate the period from August, 2009 to December, 2014.

SECONDARY OUTCOMES:
Clinical outcomes including, LDL, BP, body mass index (BMI), and cardiovascular complications. | Five years
  Baseline and 12 months for each subject; the audit cycle will be repeated annually over a period of 5 years.
Patient reported outcomes (PRO) measured by the change in SF-12v2 scores, the PEI and GRS scores at 6 months. | Five years
  Baseline and 6-month/12-month/24-month/36-month after the first administration of questionnaire.
Service utilization outcomes measured by GOPC consultation, SOPC consultation, A&E and hospital attendance rates in the past 12 months. | Five years
  Baseline and 12 months for each subject; the audit cycle will be repeated annually over a period of 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L.K. Lam, MD, Study Chair — Department of Family Medicine and Primary Care, Faculty of Medicine, The University of Hong Kong; Colman S.C. Fung, MBBS, Principal Investigator — Department of Family Medicine and Primary Care, Faculity of Medicine, The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Result] Fung CS, Chin WY, Dai DS, Kwok RL, Tsui EL, Wan YF, Wong W, Wong CK, Fong DY, Lam CL. Evaluation of the quality of care of a multi-disciplinary risk factor assessment and management programme (RAMP) for diabetic patients. BMC Fam Pract. 2012 Dec 5;13:116. doi: 10.1186/1471-2296-13-116. PMID 23216708
- [Result] Jiao FF, Fung CS, Wong CK, Wan YF, Dai D, Kwok R, Lam CL. Effects of the Multidisciplinary Risk Assessment and Management Program for Patients with Diabetes Mellitus (RAMP-DM) on biomedical outcomes, observed cardiovascular events and cardiovascular risks in primary care: a longitudinal comparative study. Cardiovasc Diabetol. 2014 Aug 21;13:127. doi: 10.1186/s12933-014-0127-6. PMID 25142791
- [Result] Jiao F, Fung CS, Wan YF, McGhee SM, Wong CK, Dai D, Kwok R, Lam CL. Long-term effects of the multidisciplinary risk assessment and management program for patients with diabetes mellitus (RAMP-DM): a population-based cohort study. Cardiovasc Diabetol. 2015 Aug 14;14:105. doi: 10.1186/s12933-015-0267-3. PMID 26268736
- [Result] Jiao F, Fung CS, Wan YF, McGhee SM, Wong CK, Dai D, Kwok R, Lam CL. Effectiveness of the multidisciplinary Risk Assessment and Management Program for Patients with Diabetes Mellitus (RAMP-DM) for diabetic microvascular complications: A population-based cohort study. Diabetes Metab. 2016 Dec;42(6):424-432. doi: 10.1016/j.diabet.2016.07.030. Epub 2016 Aug 24. PMID 27568125
- [Result] Wan EY, Fung CS, Wong CK, Choi EP, Jiao FF, Chan AK, Chan KH, Lam CL. Effectiveness of a multidisciplinary risk assessment and management programme-diabetes mellitus (RAMP-DM) on patient-reported outcomes. Endocrine. 2017 Feb;55(2):416-426. doi: 10.1007/s12020-016-1124-1. Epub 2016 Oct 3. PMID 27699706
- [Derived] Fung CS, Wan EY, Jiao F, Lam CL. Five-year change of clinical and complications profile of diabetic patients under primary care: a population-based longitudinal study on 127,977 diabetic patients. Diabetol Metab Syndr. 2015 Sep 17;7:79. doi: 10.1186/s13098-015-0072-x. eCollection 2015. PMID 26388950